CLINICAL TRIAL: NCT05178563
Title: Mechanisms of Acute Inflammation Following Periodontal Treatment (STUDENT STUDY)
Brief Title: Mechanisms of Acute Inflammation Following Periodontal Treatment
Acronym: MANTRA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRAS Project number 279840
Record Dates: First submitted 2021-11-15; First posted 2022-01-05 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Inflammation; Periodontal Diseases
MeSH Terms: conditions — Inflammation; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This study is a double blind, CONSORT-based randomized, controlled clinical trial comparing the use of local use of photodynamic therapy (PDT) pretreatment on systemic inflammation, vascular dysfunction and patient discomfort following a single session of non surgical periodontal therapy (IPT) vs. IPT alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPT+PDT (Experimental): The experimental arm consist of performing IPT in randomly assigning patients to receive local use of photodynamic therapy (PDT).
  Interventions: Procedure: IPT+PDT
- ; IPT+Placebo (Sham Comparator): This experimental arm consist of performing IPT in randomly assigning patients to receive sham use of photodynamic therapy(PDT).
  Interventions: Procedure: IPT+Placebo

INTERVENTIONS:
Procedure: IPT+PDT — The experimental arm consist of performing IPT in randomly assigning patients to receive local use of photodynamic therapy (PDT).
  Arms: IPT+PDT
Procedure: IPT+Placebo — IPT+Placebo
  Arms: ; IPT+Placebo

SUMMARY:
Periodontitis (gum disease) is a chronic inflammatory disease linked to a imbalance of oral microbiome. The most usual treatment involves removal of sub and supra-gingival plaque and calculus otherwise known as Non-surgical periodontal therapy (NSPT). Ample evidence now indicates that Periodontitis and NSPT are linked to both local and systemic inflammation. This in turn also explains the association between periodontitis and a number of systemic diseases including cardiovascular diseases.

Vascular endothelium (the innermost lining of blood vessels) exerts protective, anti-inflammatory and anti-clotting functions. As the endothelium ages, and is exposed to the damaging effects of traditional cardiovascular risk factors such as elevated blood pressure, serum cholesterol, glucose and cigarette smoking; these protective properties appear diminished, leading to a state of endothelial dysfunction (ED). Understanding the mechanisms of ED in humans could lead to new therapeutic and/or preventive strategies of CV diseases. Sufficient evidence now suggests that periodontitis and its treatment (removal of sub and supra-gingival plaque and calculus-periodontal therapy) are linked to endothelial dysfunction. Studies have extensively characterized the time-course of a single session of non surgical periodontal treatment (IPT) associated with a one week acute inflammatory response. This substantial inflammatory response is also associated with ED assessed by flow-mediated dilation (FMD) of the brachial artery at 24 hrs.

Photodynamic therapy (PDT) helps kill the local pathogens, thus preventing their systemic dissemination; which may ultimately reduce the systemic host inflammatory response generated.

DETAILED DESCRIPTION:
Periodontitis (gum disease) is a chronic inflammatory disease linked to a imbalance of oral microbiome. The most usual treatment involves removal of sub and supra-gingival plaque and calculus otherwise known as Non-surgical periodontal therapy (NSPT). Ample evidence now indicates that Periodontitis and NSPT are linked to both local and systemic inflammation. This in turn also explains the association between periodontitis and a number of systemic diseases including cardiovascular diseases.

Vascular endothelium (the innermost lining of blood vessels) exerts protective, anti-inflammatory and anti-clotting functions. As the endothelium ages, and is exposed to the damaging effects of traditional cardiovascular risk factors such as elevated blood pressure, serum cholesterol, glucose and cigarette smoking; these protective properties appear diminished, leading to a state of endothelial dysfunction (ED). Understanding the mechanisms of ED in humans could lead to new therapeutic and/or preventive strategies of CV diseases. Sufficient evidence now suggests that periodontitis and its treatment (removal of sub and supra-gingival plaque and calculus-periodontal therapy) are linked to endothelial dysfunction. Studies have extensively characterised the time-course of a single session of intense non surgical periodontal treatment (IPT) associated with a one week acute inflammatory response. This substantial inflammatory response is also associated with ED assessed by flow-mediated dilation (FMD) of the brachial artery at 24 hrs.

The efficacy of periodontal therapy is directly related to the ability of treatment to control the infection sustained by gum bacteria. Several chemical agents, such as antiseptic/bacteriostatic liquids, gels or membranes have been added to the conventional periodontal therapy with the view of improving clinical outcomes. The latest evidence advocates the use of lasers to eliminate bacteria in the periodontal pockets. Photodynamic therapy (PDT) is the process of eradication of target cells by reactive oxygen compound produced after activation of a photo-sensitiser by light of appropriate wavelength. Dental lasers used for PDT can be high-level lasers, low-level laser, and diode lasers. PDT used in dentistry for microbial killing, usually involves the use of low-intensity diode laser irradiation along with photosensitises as a means of arresting the anti-microbial activity.

Researchers and clinicians don't fully understand the mechanism underlying the local and systemic pathways involved in the role of periodontal/oral inflammation on systemic health and diseases Based on the evidence that PDT could kill the local pathogens, thus preventing their systemic dissemination; which may ultimately reduce the systemic host inflammatory response generated. The investigators hypothesized that using PDT before NSPT would result in less local and systemic inflammation/ED Understanding the mechanisms of ED in humans could lead to new beneficial and/or preventive strategies for cardio vascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female subject must be 18 years of age or over.
2. Affected by periodontitis, with at least 20 sites with PPD>4mm and have at least 20 teeth (excluding wisdom teeth).
3. Have voluntarily signed the informed consent.

Exclusion Criteria:

1. Presence of any systemic diseases (e.g., diabetes mellitus or cardiovascular, kidney, liver or lung disease).
2. Pregnant or breastfeeding.
3. Regular use of analgesic or antibiotics within 1 month before entering the study.
4. Have untreated gross carious lesions and/or insufficient restorations.
5. Allergic to any ingredient in the products provided within the trial as determined by the dental/medical professional monitoring the study.
6. Concurrent participation in other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to investigate the efficacy and safety of pre-treatment with photodynamic therapy on systemic vascular dysfunction (assessed via FMD) following a single session of non-surgical periodontal therapy (IPT) vs. IPT alone. | 24 hours post op
  The primary outcome -Flow-mediated dilatation (an ultra-sound scan) of the brachial artery- at 24 hours between study groups to see changes in vessel wall elasticity.
  Vessel Wall Elasticity (Vascular dysfunction) will be observed in the population of periodontitis patients who will undergo IPT with or without photodynamic therapy, using Flow mediated dilatation (FMD) which is an ultra-sound scan of brachial artery (before and after treatment).
  FMD measurements will be done to assess the % change in vessel wall diameter.

SECONDARY OUTCOMES:
FMD at different time points following treatment between study groups. | 0, 1, 3, 7 and 180 days following treatment.
  FMD at 0,1, 3, 7 and 180 days following treatment between study groups. FMD measurements will be done to assess the % change in vessel wall diameter.
Pulse wave velocity (PWV) at different time points following treatment between study groups. | 0, 1, 3, 7 and 180 days following treatment.
  PWV at 0,1, 3, 7 and 180 days following treatment between study groups. Pulse wave velocity (PWV) is a measure of arterial stiffness between to measurement sites . PWV is measured according to pulse rate detected.
Evaluate the effect of PDT /IPT on biomarkers of systemic inflammation. | 0, 1, 3, 7 and 180 days following treatment.
  Evaluate the effect of PDT /IPT on acute phase biomarkers of systemic inflammation (hs-CRP, Serum amyloid A (SAA).
  The values for biomarkers hs-CRP and SAA-mg/L,will be expressed in mg/L
  The effect will be determined by changes in units of measurement for each blood marker as applicable.
Evaluate the effect of PDT /IPT on biomarkers of systemic inflammation. | 0, 1, 3, 7 and 180 days following treatment.
  Evaluate the effect of PDT /IPT on cellular adhesion molecule biomarkers of systemic inflammation comprising of (ICAM-1, VCAM-1)
  The values forICAM-1 and VCAM-1 will be expressed in ng/mL
  The effect will be determined by changes in units of measurement for each blood marker as applicable.
Evaluate the effect of PDT /IPT on biomarkers of systemic inflammation. | 0, 1, 3, 7 and 180 days following treatment.
  Evaluate the effect of PDT /IPT on cytokine biomarkers of systemic inflammation which are Interleukins (IL-6, IL-8, IL-10, IL-17A, IL-18, IL-23), Interferon (IFN- γ), Tumour necrosis factor (TNF-α), Monocyte chemotactic protein (MCP-1) and Thrombopoeitin (TPO)
  The values for all these cytokines comprising of Interleukins(IL)- IL-6, IL-8, IL-10, IL-17A, IL-18, IL-23 will be expressed in pg/ml.
  The value of IFN- γ-will be expressed in pg/ml.
  The value of TNF-α will be expressed in pg/ml.
  The value of MCP-1 will be expressed in pg/ml.
  The value of TPO will be expressed in pg/ml.
  The effect will be determined by changes in units of measurement for each cytokine blood marker which will be expressed in pg/ml for all these markers.
Evaluate the effect of PDT /IPT on biomarkers of systemic inflammation. | 0, 1, 3, 7 and 180 days following treatment.
  Evaluate the effect of PDT /IPT on lipid biomarkers of systemic inflammation- lipidemic markers comprising of HDL, LDL, TG.
  The values for all lipidemic markers will be expressed as:
  HDL-as mg/dL, LDL-mg/dL, TG- mmol/L
  The effect will be determined by changes in units of measurement for each blood marker as applicable.
Evaluate the effect of PDT /IPT on markers of endothelial function | 0, 1, 3, 7 and 180 days following treatment.
  Evaluate the effect of PDT /IPT on markers of endothelial activation (E-Selectin, ICAM-3, P-Selectin, Thrombomodulin) at different time points following treatment between study groups.
  The value of these biomarkers will be expressed as E-Selectin- pg/ml, ICAM-3-ng/mL, P-Selectin- pg/ml, Thrombomodulin- pg/ml.
  The effect will be determined by changes in units of measurement for each blood marker as applicable.
Evaluate the effect of PDT /IPT on glycemic profile | 0, 1, 3, 7 and 180 days following treatment.
  Evaluate the effect of PDT /IPT on glycemic profile at different time points following treatment between study groups.
  Glycemic values will be measured as blood glucose levels are measured in units called mmol/L (pronounced milli-moles-per-litre).
Evaluate the effect of PDT /IPT on oxidative profile | 0, 1, 3, 7 and 180 days following treatment.
  Evaluate the effect of PDT /IPT on oxidative profile (d-ROMs) at different time points following treatment between study groups.
  Oxidative profile (d-ROMs) will be measured in Carratelli units..
Evaluate the effect of PDT/IPT on the monocyte subset, monocyte platelet aggregate (MPA) , and circulating endothelial progenitor cells (EPC). | 0, 1, 3, 7 and 180 days following treatment.
  Evaluate the effect of PDT/IPT on the monocyte subset, monocyte platelet aggregate (MPA) , and circulating endothelial progenitor cells (EPC) assessed via flow cytometry in a population of patients suffering from periodontitis at different time points following treatment between study groups. The values will be determined by changes in cell count over time.
Investigate the periodontal clinical parameters following IPT with and without the use of PDT. | 6 months post intervention
  Clinical periodontal parameters differences at following PDT+IPT or IPT. Clinical periodontal parameters will be recorded by a single calibrated examiner using a manual University of North Carolina (UNC-15) periodontal probe to see level of gingival margin with reference to a fixed point on the tooth (cementoenamel junction(CEJ)). The measurements will be recorded in millimetres.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastman Dental Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No